CLINICAL TRIAL: NCT02858258
Title: Autologous Transplantation After a Rituximab/Ibrutinib/Ara-c Containing iNduction in Generalized Mantle Cell Lymphoma - a Randomized European Mcl Network Trial
Brief Title: ASCT After a Rituximab/Ibrutinib/Ara-c Containing iNduction in Generalized Mantle Cell Lymphoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Prof. Dr. M. Dreyling (co-chairman) (Other)
Collaborators: LMU Klinikum (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. M. Dreyling (co-chairman), Sponsor Delegated Person / Coordinating Prinicipal Investigator, European Mantle Cell Lymphoma Network
Organization: European Mantle Cell Lymphoma Network (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRIANGLE
Record Dates: First submitted 2016-07-14; First posted 2016-08-08 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Mantle Cell Lymphoma
Keywords: MCL
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Rituximab; ibrutinib; Neoadjuvant Therapy; Tromethamine; Maintenance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Standard Arm A (Active Comparator): R-CHOP/R-DHAP: Alternating 3 cycles of R-CHOP in cycle 1,3,5 and 3 cyles of R-DHAP in cycle 2,4,6; each 21 day cycle
  Drug: R-CHOP/R-DHAP
  ASCT conditioning (ASCT: autologous stemm cell transplantation) Drug: THAM or BEAM
  Interventions: Drug: R-CHOP/R-DHAP; Drug: ASCT conditioning
- Experimental Arm A+I (Experimental): R-CHOP+Ibrutinib/R-DHAP: Alternating 3 cycles of R-CHOP + Ibrutinib at Days 1-19 in cycle 1,3,5 and 3 cyles of R-DHAP in cycle 2,4,6; each 21 day cycle
  Drug: R-CHOP/R-DHAP Drug: Ibrutinib (Induction)
  ASCT conditioning (ASCT: autologous stemm cell transplantation) Drug: THAM or BEAM
  2 years Ibrutinib Maintenance Drug: Ibrutinib (Maintenace)
  Interventions: Drug: R-CHOP/R-DHAP; Drug: Ibrutinib (Induction); Drug: ASCT conditioning; Drug: Ibrutinib (Maintenance)
- Experimental Arm I (Experimental): R-CHOP+Ibrutinib / R-DHAP: Alternating 3 cycles of R-CHOP + Ibrutinib at Days1-19 in cycle 1,3,5 and 3 cyles of R-DHAP in cycle 2,4,6; each 21 day cycle
  Drug: R-CHOP/R-DHAP Drug: Ibrutinib (Induction)
  2 years Ibrutinib Maintenance Drug: Ibrutinib (Maintenance)
  Interventions: Drug: R-CHOP/R-DHAP; Drug: Ibrutinib (Induction); Drug: Ibrutinib (Maintenance)

INTERVENTIONS:
Drug: R-CHOP/R-DHAP — Drug: R-CHOP/DHAP Alternating 3x R-CHOP (Rituximab , Cyclophosphamide ,Doxorubicine ,Vincristine , Prednisone) / 3x R-DHAP (Rituximab , Dexamethasone, Ara-C, Cisplatine, G-CSF)
  Other Names: rituximab, CHOP, DHAP
Drug: Ibrutinib (Induction) — Ibrutinib: only in cycle 1,3,5 on Day 1-19
  Other Names: Imbruvica
  Arms: Experimental Arm A+I; Experimental Arm I
Drug: ASCT conditioning — ASCT conditioning THAM or BEAM, stratified per site before trial activation at site
  THAM (TBI (total body irradiation), Ara-C, Melphalan) or
  BEAM (BCNU, Etoposide, Cytarabine, Melphalan)
  Other Names: THAM or BEAM
  Arms: Experimental Arm A+I; Standard Arm A
Drug: Ibrutinib (Maintenance) — Ibrutinib (Maintenance), daily 560 mg for 2 years;
  Other Names: Imbruvica
  Arms: Experimental Arm A+I; Experimental Arm I

SUMMARY:
The primary objective of the the trial is to establish one of three study arms, as future standard based on the comparison of the investigator-assessed failure-free survival.

DETAILED DESCRIPTION:
Objectives and Endpoints

Primary Objective:

To establish one of three study arms, R-CHOP/R-DHAP followed by ASCT (control arm A), R-CHOP+ibrutinib /R-DHAP followed by ASCT and ibrutinib maintenance experimental arm A+I), and R-CHOP+ibrutinib /R-DHAP followed by ibrutinib maintenance experimental arm I) as future standard based on the comparison of the investigator-assessed failure-free survival (FFS).

Secondary Objectives:

* To compare the efficacy of the three treatment arms in terms of secondary efficacy endpoints
* To determine the safety and tolerability of ibrutinib during induction immuno-chemotherapy and during maintenance and to compare the safety profile of the three treatment arms in terms of secondary toxicity endpoints

Primary Endpoint:

FFS defined as time from start of treatment to stable disease at end of immuno-chemotherapy, progressive disease, or death from any cause.

Secondary Efficacy Endpoints:

* Overall survival (OS)
* Progression-free survival (PFS) from randomization, from end of induction immuno-chemotherapy in patients with CR or PR at end of induction immuno-chemotherapy, and from the staging 6 weeks after end of induction assessment (at month 6)
* Overall response and complete remission rates at midterm, at end of induction, 3 months after end of induction immunochemotherapy (at month 6)
* PR to CR conversion rate during follow-up after end of induction immuno-chemotherapy

Secondary Toxicity Endpoints:

* Rates of AEs, SAEs, and SUSARs by CTC grade (Version 4.03) during induction immuno-chemotherapy and during periods of follow-up after response to immune-chemotherapy
* Cumulative incidence rates of SPMs

Exploratory Objectives:

* To compare feasibility of ASCT in arm A+I vs. arm A
* To compare minimal residual disease status between the three treatment groups
* To determine the impact of ibrutinib during induction immuno-chemotherapy and during maintenance therapy on the minimal residual disease status
* To determine the prognostic value of minimal residual disease status
* To determine the prognostic value of positron emission tomography with fluorine 18-fluorodeoxyglucose
* To determine clinical and biological prognostic and predictive factors
* To determine the role of total body irradiation (TBI) in ASCT conditioning

Exploratory Endpoints:

* Rate of successful stem cell mobilisations (success: separation of at least 2x2x10(6) CD34-positive cells, including a back-up)
* Rate of molecular remissions (MRD-negative patients) at midterm, at end of induction immuno-chemotherapy, and at staging time-points during follow-up in patients with remission after end of induction immuno-chemotherapy
* Time to molecular remission from start of therapy
* Time to molecular relapse for patients in clinical and molecular remission after end of induction immunochemotherapy
* RD in FDG-PET negative or positive patients after induction and ASCT

Exploratory objectives may be evaluated only in a subset of patients according to local standards and resources.

ELIGIBILITY:
Inclusion Criteria:

All patients must meet the following criteria:

* Histologically confirmed diagnosis of MCL according to WHO classification
* suitable for high-dose treatment including high-dose Ara-C
* Stage II-IV (Ann Arbor)
* Age ≥ 18 years and ≤ 65 years
* Previously untreated MCL
* At least 1 measurable lesion; in case of bone marrow infiltration only, bone marrow aspiration and biopsy is mandatory for all staging evaluations.
* ECOG/WHO performance status ≤ 2
* The following laboratory values at screening (unless related to MCL):

  * Absolute neutrophil count (ANC) ≥1000 cells/µL
  * Platelets ≥100,000 cells/µL
  * Transaminases (AST and ALT) ≤3 x upper limit of normal (ULN)
  * Total bilirubin ≤2 x ULN unless due to known Morbus Meulengracht [Gilbert-Meulengracht-Syndrome])
  * Creatinine ≤2 mg/dL or calculated creatinine clearance ≥ 50 mL/min
* Written informed consent form according to ICH/EU GCP and national regulations
* Sexually active men and women of child-bearing potential must agree to use highly effective contraceptives (eg, condoms, implants, injectables, combined oral contraceptives, intrauterine devices, sexual abstinence, or sterilized partner) while on study; this should be maintained for 90 days after the last dose of study drug.

Exclusion Criteria:

Any potential subject who meets any of the following criteria will be excluded from participating in the study.

* Major surgery within 4 weeks prior to randomization.
* Requires anticoagulation with warfarin or equivalent vitamin K antagonists (eg phenprocoumon).
* History of stroke or intracranial hemorrhage within 6 months prior to randomization.
* Requires treatment with strong CYP3A4/5 inhibitors.
* Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of ibrutinib capsules, or put the study outcomes at undue risk.
* Vaccinated with live, attenuated vaccines within 4 weeks prior to randomization.
* Known CNS involvement of MCL
* Clinically significant hypersensitivity (eg, anaphylactic or anaphylactoid reactions to the compound of ibrutinib itself or to the excipients in its formulation)
* Known anti-murine antibody (HAMA) reactivity or known hypersensitivity to murine antibodies
* Previous lymphoma therapy with radiation, cytostatic drugs, anti-CD20 antibody or interferon except prephase therapy according to trial protocol
* Serious concomitant disease interfering with a regular therapy according to the study protocol:

  * Cardiac (Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of Screening, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification or LVEF below LLN )
  * Pulmonary (e.g. chronic lung disease with hypoxemia)
  * Endocrinological (e.g. severe, not sufficiently controlled diabetes mellitus)
  * Renal insufficiency (unless caused by the lymphoma): creatinine > 2x normal value and/or creatinin clearance < 50 ml/min)
  * Impairment of liver function (unless caused by the lymphoma): transaminases > 3x normal or bilirubin > 2,0 mg/dl unless due to morbus Meulengracht (Gilbert-Meulengracht-Syndrome)
* Patients with unresolved hepatitis B or C infection or known HIV positive infection (mandatory test)
* Prior organ, bone marrow or peripheral blood stem cell transplantation
* Concomitant or previous malignancies within the last 3 years other than basal cell skin cancer or in situ uterine cervix cancer
* Pregnancy or lactation
* Any psychological, familiar, sociological, or geographical condition potentially hampering compliance with the study protocol and follow up schedule
* Subjects not able to give consent
* Subjects without legal capacity who are unable to understand the nature, scope, significance and consequences of this clinical trial
* Participation in another clinical trial within 30 days before randomization in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 870 (Estimated)
Dates: Start 2016-07; Primary Completion 2021-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Failure Free Survival | From start of treatment until stable disease at end of immuno-chemotherapy, progressive disease, or death from any cause, whichever comes first, assessed up to 120 months.

SECONDARY OUTCOMES:
Overall Survival | From start of treatment until the date of first documented progression, assessed up to 120 months.
Number of participants with treatment-related adverse events as assessed by CTC Version 4.03 | From start of Ibrutinib treatment during induction immuno-chemotherapy and during maintenance and to compare the safety profile of the three treatment arms in terms of secondary toxicity endpoints. Through study conduction, an average of up to 30 months.
  Safety and tolerability
Progression-free survival (PFS) | PFS is the time to progression or death from any cause. Assed up to 120 months.
Number of Secondary Primary Malignancies | From start of treatment through the study conduction, up to 120 months.
  Toxicity Endpoints
Number of Adverse Events by CTC grade (Version 4.03) | From start of treatment through the study conduction, up to 120 months.
  Toxicity Endpoints

CONTACTS AND LOCATIONS:
Overall Officials: Martin Dreyling, Prof., Principal Investigator — Klinikum der Universität München
Locations (112):
- Denmark (6):
  - Aalborg University Hospital, Dept of Hematology, Aalborg
  - Aarhus University Hospital, Dept of Hematology, Aarhus C
  - Rigshospitalet, Clinic of Hematology, Copenhagen
  - Herlev Hospital, Department of Hematology L121, Herlev
  - Odense University Hospital, Dept of Hematology X, Odense C
  - Sjaelland University Hospital, Dept of Hematology, Roskilde
- Germany (60):
  - Zentralklinik Augsburg, II. Med. Klinik, Hämatologie int. Onkologie, Augsburg
  - Onkologische Gemeinschaftspraxis Dr. Janssen/Dr. Reichert in der Ubbo-Emmius-Klinik, Aurich
  - Klinikum Bayreuth, Klinik f. Onkologie und Hämatologie, Bayreuth
  - Vivantes Klinikum Am Urban, Klinik f. Innere Medizin, Hämatologie und Onkologie, Berlin
  - Charité Univ.-Medizin Berlin, Med. Klinik - Hämatologie, Onkologie und Tumorimmunologie, Berlin
  - Helios Klinikum Berlin-Buch, Hämatologie, Onkologie und Tumorimmunologie, Berlin
  - Knappschaftskrankenhaus Bochum-Langendreer, Bochum
  - Universitätsklinikum Bonn, Bonn
  - Diako ev. Diakonie-KH gGmbH, Med. Klinik II, Hämatologie und Onkologie, Bremen
  - Klinikum Chemnitz gGmbH, Klinik f. Innere Medizin II, Chemnitz
  - Uniklinik Köln, Klinik I für Innere Medizin, Cologne
  - DONAUISAR Klinikum Deggendorf, Innere Medizin II, Deggendorf
  - St.-Johannes-Hospital, Dortmund
  - Gemeinschaftspraxis Dr. Mohm und Prange-Krex - Fachärzte für Innere Medizin und Hämatologie und Onkologie, Dresden
  - Universitätsklinikum Carl Gustav Carus an der Technischen Universität Dresden, Dresden
  - Universitätsklinikum Düsseldorf, Klinik f. Hämatologie, Onkologie und klinische Immunologie, Düsseldorf
  - Marien Hospital Düsseldorf, Düsseldorf
  - Helios Klinikum Erfurt GmbH, Zentrum f. Innere Medizin u. internistische Onkologie, Hämostaseologie, Erfurt
  - Universitätsklinikum Erlangen, Med. Klinik 5, Hämatologie und internistische Onkologie, Erlangen
  - St.-Antonius-Hospital Eschweiler, Klinik für Hämatologie und Onkologie, Eschweiler
  - Universitätsklinikum Essen, Klinik f. Hämatologie, Essen
  - Universitätsklinikum Freiburg, Klinik f. Innere Medizin, Hämatologie, Onkologie u. Stammzelltransplantation, Freiburg im Breisgau
  - Universitätsmedizin Göttingen, Zentrum f. Innere Medizin, Klinik f. Hämatologie und Medizinische Onkologie, Göttingen
  - Universitätsmedizin Greifswald, Klinik u. Poliklinik f. Innere Medizin C, Hämatologie u. Onkologie-, Transplantationszentrum, Greifswald
  - Katholisches Krankenhaus Hagen gGmbH, St.-Marien-Hospital, Klinik f. Hämatologie und Onkologie, Hagen
  - Universitätsklinikum Hamburg-Eppendorf (UKE), II. Med. Klinik u. Poliklinik, Onkologie, Hämatologie, KMT, Hamburg
  - Asklepios Klinik Altona, II. Med.Abt. f. Hämatologie und internistische Onkologie, Stammzelltransplantation, Hamburg
  - Universitätsklinikum Heidelberg, Med. Klinik - Innere Medizin V - Hämatologie, Onkologie und Rheumatologie, Heidelberg
  - Universitätsklinikum des Saarlandes, Klinik f. Innere Medizin I Hämatologie & Onkologie, Homburg
  - Klinikum Idar-Oberstein GmbH, Medizinische Klinik I, Idar-Oberstein
  - Universitätsmedizin Jena, Klinik f. Innere Medizin II, Abteilung Hämatologie u. Internistische Onkologie, Jena
  - Städtisches Klinikum Karlsruhe, Med. Klinik III, Hämatologie und Onkologie, Karlsruhe
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel, Klinik f. Innere Medizin II - Hämatologie und Onkologie, Kiel
  - Gemeinschaftsklinikum Mittelrhein gGmbH, Ev. Stift St. Martin, Klinik f. Innere Medizin, Koblenz
  - Praxisklinik f. Hämatologie und Onkologie Koblenz, Koblenz
  - Onkologisch-Hämatologische Praxis Dr. Vehling-Kaiser, Landshut
  - Klinikum Landshut gGmbH, Med. Klinik III, Hämatologie/Internistische Onkologie, Landshut
  - Caritas-KHLebach, Gemeinschaftspraxis f. Hämatologie und Onkologie, Onkologisches Zentrum Lebach, Lebach
  - Universitätsklinikum Leipzig AöR, selbständige Abteilung f. Hämatologie und Internistische Onkologie, Hämostaseologische Ambulanz, Leipzig
  - Klinikum Lippe GmbH, Onkologie und Hämatologie, Lemgo
  - Klinikum der Stadt Ludwigshafen am Rhein gGmbH, Med. Klinik A, Ludwigshafen
  - Universitätsklinikum Magdeburg AöR, Klinik f. Hämatologie und Onkologie, Magdeburg
  - Universitätsmedizin der Univ. Mainz, III. Med. Klinik u. Poliklinik, Mainz
  - Johannes Wiesling Klinikum Minden, Klinik f. Hämatologie/Onkologie, Hämostaseologie und Palliativmedizin, Minden
  - Klinikum der Universität München, Med. Klinik und Poliklinik III, München
  - Klinikum Rechts der Isar, III. Med. Klinik - Hämatologie und Onkologie, München
  - Universitätsklinikum Münster, Med. Klinik A, Translationale Onkologie / Lymphome, Münster
  - Klinikum Nürnberg,5. Medizinische Klinik, Onkologie / Hämatologie, Nuremberg
  - Klinikum Oldenburg gGmbH, Med. Klinik II, Oldenburg
  - Klinikum Ernst von Bergmann Potsdam gGmbH, Zentrum f. Innere Medizin, Klinik f. Hämatologie und Onkologie, Potsdam
  - KH Barmherzige Brüder, Klinik f. Onkologie und Hämatologie, Regensburg
  - Universitätsmedizin Rostock, Abt. f. Hämatologie und Onkologie, Klinik und Poliklinik für Innere Medizin, Rostock
  - Klinikum Stuttgart - Katharinenhospital, Klinik f. Hämatologie und Onkologie, Stuttgart
  - Robert-Bosch-Krankenhaus, Abt.f. Hämatologie und Onkologie, Stuttgart
  - Klinikum Traunstein, Hämatologie - Onkologie- Palliativmedizin, Traunstein
  - Klinikum Mutterhaus der Borromäerinnen gGmbH, Okologisches Zentrum, Trier
  - Universitätsklinikum Tübingen, Med Klinik I, Innere Medizin II, Tübingen
  - Universitätsklinikum Ulm, Klinik für Innere Medizin III, Ulm
  - Klinikum Wolfsburg, Med. Klinik II, Wolfsburg
  - Universitätsklinikum Würzburg, Med. Klinik u. Poliklinik II /ZIM, Würzburg
- Italy (33):
  - Azienda Ospedaliera SS. Antonio e Biagio e C. Arrigo, SC Ematologia, Alessandria
  - Policlinico S. Orsola Malpighi, Istituto di Ematologia e Oncologia Medica Seragnoli, Bologna
  - Comprensorio Sanitario di Bolzano, Ematologia e trapianto di midollo osseo, Bolzano
  - Spedali Civili, Struttura Complessa di Ematologia, Brescia
  - Ospedale Businco, UO Ematologia - CTMO, Cagliari
  - ASO S. Croce e Carle, S.C. di Ematologia e Trapianto di Midollo Osseo, Cuneo
  - AOU Policlinico Careggi, Unità Funzionale di Ematologia, Florence
  - IRCCS AOU S. Martino - IST, Clinica Ematologia, Genova
  - IRCCS AOU S. Martino - IST, Ematologia, Genova
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Ematologia, Meldola (FC)
  - Istituto Scientifico San Raffaele, Unità Ricerca Clinica Linfomi, Milan
  - Ospedale Niguarda, Struttura Complessa di Ematologia, Milan
  - Università di Modena e Reggio Emilia Policlinico - COM Centro Oncologico Modenese, Dipartimento di Oncologia ed Ematologia, Modena
  - Ospedale S. Gerardo, Divisione di Ematologia, Monza
  - "IRCCS Istituto Nazionale dei Tumori di Napoli - Pascale", Ematologia Oncologica, Napoli
  - AOU Maggiore della Carità - Università del Piemonte Orientale, S.C.D.U Ematologia, Novara
  - AO Ospedali Riuniti Villa Sofia-Cervello, Divisione di Ematologia, Palermo
  - IRCCS Fondazione Policlinico San Matteo, Clinica Ematologia, Pavia
  - Azienda Ospedaliera Pisana Ospedale "S.Chiara", Dipartimento di Oncologia Divisione di Ematologia, Pisa
  - Ospedale S. Maria delle Croci, U.O di Ematologia, Ravenna
  - Azienda Ospedaliera Bianchi, Melacrino, Morelli, Divisione di Ematologia, Reggio Calabria
  - Azienda Ospedaliera Arcispedale Santa Maria Nuova - IRCCS, Ematologia, Reggio Emilia
  - Ospedale degli Infermi, U.O. Ematologia, Rimini
  - Policlinico Tor Vergata, UOC Oncoematologia, Roma
  - Università La Sapienza, Ematologia, Roma
  - Casa Sollievo della Sofferenza, U.O. Ematologia, San Giovanni Rotondo
  - A.O. Città della Salute e della Scienza, SC Ematologia, Torino
  - A.O. U. Città della Salute e della Scienza, S C Ematologia U, Torino
  - Ospedale Cà Foncello, U.O.C. Ematologia, Treviso
  - Ospedale Cardinale Panico, Divisione di Ematologia, Tricase
  - ASUI Integrata di Udine, Clinica Ematologia, Udine
  - Ospedale Policlinico G.B. Rossi, "Centro trapianto midollo osseo Ematologia", Verona
  - Ospedale S. Bortolo, Ematologia, Vicenza
- Norway (5):
  - Haukeland University Hospital , Dept. of Oncology and Medical Physics, Bergen
  - Oslo University Hospital, Dept of Oncology, Oslo
  - Stavanger University Hospital, Division for Hematology&Oncology, Stavanger
  - UNN Tromsø, Oncology Dep, Tromsø
  - St. Olavs Hospital, Department of Oncology, Trondheim
- Sweden (8):
  - Sahlgrenska University Hospital, Section of Hematology and Coagulation, Dept of internal medicine, Gothenburg
  - University Hospital, Dept of Hematolgy, Linköping
  - Sunderbyn Hospital, Dept of Medicine, Luleå
  - Skane University Hospital, Lund
  - Örebro University Hospital, Dept of Oncology, Örebro
  - Karolinska University Hospital, Center of Hematology, Stockholm
  - Norrland University Hospital, Dept of Oncology, Umeå
  - Academic Hospital, Dept of Oncology, Uppsala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dreyling M, Doorduijn J, Gine E, Jerkeman M, Walewski J, Hutchings M, Mey U, Riise J, Trneny M, Vergote V, Shpilberg O, Gomes da Silva M, Leppa S, Jiang L, Stilgenbauer S, Kerkhoff A, Jachimowicz RD, Celli M, Hess G, Arcaini L, Visco C, van Meerten T, Wirths S, Zinzani PL, Novak U, Herhaus P, Benedetti F, Sonnevi K, Hanoun C, Hanel M, Dierlamm J, Pott C, Klapper W, Gozel D, Schmidt C, Unterhalt M, Ladetto M, Hoster E. Ibrutinib combined with immunochemotherapy with or without autologous stem-cell transplantation versus immunochemotherapy and autologous stem-cell transplantation in previously untreated patients with mantle cell lymphoma (TRIANGLE): a three-arm, randomised, open-label, phase 3 superiority trial of the European Mantle Cell Lymphoma Network. Lancet. 2024 May 25;403(10441):2293-2306. doi: 10.1016/S0140-6736(24)00184-3. Epub 2024 May 2. PMID 38705160
- [Derived] Kumar A. What is the role of up-front autologous stem cell transplantation in mantle cell lymphoma? Hematology Am Soc Hematol Educ Program. 2022 Dec 9;2022(1):155-162. doi: 10.1182/hematology.2022000333. PMID 36485104